CLINICAL TRIAL: NCT02137135
Title: The Influence of the Menstrual Cycle on Acute and Persistent Pain After Laparoscopic Cholecystectomy
Brief Title: Menstrual Phase and Postoperative Pain
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, SINEM SARI, MD, Assistant Professor, Aydin Adnan Menderes University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SARI-05
Record Dates: First submitted 2014-05-12; First posted 2014-05-13 (Estimated); Last update posted 2014-05-13 (Estimated); Status verified 2014-05

CONDITIONS: Acute Postoperative Pain; Chronic Postoperative Pain
Keywords: chronic postoperative pain; menstrual cycle
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- follicular phase (Experimental): Visual anlogue score vas used to evaluate pain. The anxiety/depression scale (HAD) was used to assess anxiety and depression. The SF 12 test (SHORT FORM 12) was used to evaluate quality of life.
  Interventions: Other: HAD scale; Other: The SF 12 test; Other: Visual analogue score
- luteal phase (Active Comparator): Visual anlogue score vas used to evaluate pain. The anxiety/depression scale (HAD) was used to assess anxiety and depression. The SF 12 test (SHORT FORM 12) was used to evaluate quality of life.
  Interventions: Other: HAD scale; Other: The SF 12 test; Other: Visual analogue score

INTERVENTIONS:
Other: HAD scale — The anxiety/depression scale (HAD) was used to assess anxiety and depression.
  Other Names: The anxiety/depression scale
Other: The SF 12 test — The SF 12 test (SHORT FORM 12) was used to evaluate quality of life.
  Other Names: SHORT FORM 12
Other: Visual analogue score — Visual analogue score vas used to evaluate pain.
  Other Names: VAS score

SUMMARY:
Fluctuations of female sex hormones during the menstrual cycle influence pain perception. Endogenous pain is pronounced in the follicular phase of the menstrual cycle. The investigators tested the primary hypothesis that the women having surgery during their follicular phase have more acute pain and require more opioids than those in the luteal phase, and secondarily the investigators tested that women who have surgery during their follicular phase have more incisional pain at 3 month postoperatively.

DETAILED DESCRIPTION:
127 adult females having laparoscopic cholecystectomy were randomized to have surgery during the luteal or follicular phase of their menstrual cycle. Standardized anesthesia and pain management regimen was given to all patients. Pain and analgesic consumption were evaluated in PACU and every four hours in first 24 hours. Adverse effects were also questioned every four hours. Time to oral intake and ambulation were recorded. Post-surgical pain, hospital anxiety and depression scale, and SF-12 questionnaire were also evaluated at 1- and 3-month visits.

ELIGIBILITY:
Inclusion Criteria:

* Women with a negative urine pregnancy test

Exclusion Criteria:

* Patients with pre-existing pain syndromes
* Patients using routinely using opioids
* Patients using hormone preparations in the last 6 months
* Patients with hysterectomy
* Patients breastfeeding in the previous 6 months
* Patients with body mass index >35 kg/m2

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2012-08; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Persistent surgical pain after laparoscopic cholecystectomy assessed by VAS scale | 3 months

SECONDARY OUTCOMES:
The anxiety and depression was evaluated with Hospital anxiety and depression scale. | 3 months

OTHER OUTCOMES:
Quality of life was evaluated with SF 12 test. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Betul Kozanhan, Specialist Doctor, Principal Investigator — Konya Education and Research Hospital, Anesthesiology and Reanimation Department, Konya; Turkey; Ayse Ilksen Egilmez, Specialist Doctor, Principal Investigator — Konya Education and Research Hospital, Anesthesiology and Reanimation Department, Konya; Turkey; Aykut Soyder, Assistant Professor, Principal Investigator — Adnan Menderes University Medical Faculty, General Surgery Department, Aydin; Turkey; Fabrizio Galimberti, Medical Student, Principal Investigator — Cleveland ClinicLernerCollege of Medicine, Cleveland, Ohio; Daniel I. Sessler, Professor and Ch, Principal Investigator — Department of Outcomes Research, Cleveland Clinic; Alparslan Turan, Associate Professor, Principal Investigator — Associate Professor of Anesthesiology, Department of Outcomes Research, Cleveland Clinic; Osman Nuri Aydın, Professor, Principal Investigator — Adnan Menderes University Medical Faculty, Anesthesiology and Reanimation Department, Aydin; Turkey
Locations (1):
- Adnan Menderes University Medical Faculty, Anesthesiology and Reanimation Department, Aydin, Turkey (Türkiye)

REFERENCES:
- [Result] Kuba T, Quinones-Jenab V. The role of female gonadal hormones in behavioral sex differences in persistent and chronic pain: clinical versus preclinical studies. Brain Res Bull. 2005 Aug 15;66(3):179-88. doi: 10.1016/j.brainresbull.2005.05.009. PMID 16023915